CLINICAL TRIAL: NCT01459770
Title: Medication Intervention in Transitional Care to Optimize Outcomes & Costs in CKD & ESRD
Brief Title: Medication Intervention in Transitional Care to Optimize Outcomes & Costs for CKD & ESRD
Acronym: CKD/ESRD-MIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Medical Research Center (Other)
Collaborators: Washington State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Health Sciences & Services Authority of Spokane County (Unknown); Providence Sacred Heart Medical Center & Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34DK094016-01 (NIH); R34DK094016-01 (NIH); RFP # 7 (Other Grant/Funding Number: Washington State Health Sciences & Services Authority)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
Keywords: glomerular filtration rate; albuminuria; medical therapy; hospital discharge; hospital readmission; CKD complications; CKD risk factors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Albuminuria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): usual care for hospital discharge:
  1. CKD group
  2. ESRD group
  Interventions: Other: Usual care for hospital discharge
- intervention (Active Comparator): pharmacist administered medication information transfer intervention
  1. CKD group
  2. ESRD group
  Interventions: Other: Medication Information Transfer Intervention

INTERVENTIONS:
Other: Medication Information Transfer Intervention — A pharmacist will visit participants randomized to the intervention group in their homes within 5 days of hospital discharge to administer the 5As Medication Self-Management intervention: Assessment, Advise, Agreement, Assistance, Arrangements.
  Arms: intervention
Other: Usual care for hospital discharge — Patients will receive medication information according to standard practice for discharge of hospitalized patients.
  Arms: control

SUMMARY:
Transitional care strategies focused on enhancing the accuracy and comprehensiveness of medication information transfer will lead to improved health outcomes among hospitalized patients with chronic kidney disease.

DETAILED DESCRIPTION:
Patients with CKD and ESRD have more co-morbidities, are hospitalized more often and for longer lengths of stay, and incur greater healthcare costs than patients with other chronic conditions. Enhanced hospital to home transitional care interventions have been shown to improve medication information transfer, reduce hospital readmissions, and slow the progression of declining health in the general population of hospitalized patients. What is not known is the impact enhanced transitional care can have for a very high-risk population, such as those with CKD and ESRD. Interventions that prevent or slow CKD progression, i.e. blood pressure control and intensive glycemic control in patients with diabetes, are all highly dependent on meticulous medication management.

For hospitalized patients with CKD or ESRD who are transitioning to home, accurate and comprehensive information transfer is essential to optimal medication management. CKD and ESRD patients are in critical need of improved transitional care that includes accurate and comprehensive medication information transfer. The main objective of this application is to pilot-test the effectiveness of a medication information transfer intervention to improve clinically-relevant outcomes. To this end, the following Specific Aims will be achieved: 1. Evaluate the impact of transitional care interventions on acute care utilization following hospital discharge among patients with CKD or ESRD. 2. Evaluate the impact of transitional care strategies on management of CKD or ESRD management and complications.

ELIGIBILITY:
Inclusion Criteria for CKD arm:

1. Hospitalized patients
2. > 21 years of age
3. Diagnosis of CKD stages 3-5, not treated by dialysis

Inclusion Criteria for ESRD arm:

1. Hospitalized patients
2. > 21 years of age
3. Patients treated with hemodialysis or peritoneal dialysis

Exclusion Criteria:

1. Kidney Transplant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
acute care utilization | 90 days
  Acute care utilization defined by emergency department visits and hospitalizations in the first 30 and 90 days after discharge from the index hospitalization.

SECONDARY OUTCOMES:
CKD status, risk factors and complications | 30 and 90 days
  blood pressure, eGFR, urine albumin/creatinine ratio, fasting glucose, HbA1c (in the diabetic subgroup), lipids, hemoglobin, phosphorus, PTH, serum potassium.
ESRD status, risk factors and complications: | 30 and 90 days
  blood pressure, fasting glucose,HbA1c (in the diabetic subgroup), lipids, hemoglobin, phosphorus, PTH, serum potassium

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R Tuttle, MD, Principal Investigator — Providence Sacred Heart Medical Center and Children's Hospital; University of Washington School of Medicine; Cynthia L Corbett, PhD, Principal Investigator — Washington State University College of Nursing
Locations (1):
- Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alicic RZ, Short RA, Corbett CL, Neumiller JJ, Gates BJ, Daratha KB, Barbosa-Leiker C, McPherson S, Chaytor NS, Dieter BP, Setter SM, Tuttle KR. Medication Intervention for Chronic Kidney Disease Patients Transitioning from Hospital to Home: Study Design and Baseline Characteristics. Am J Nephrol. 2016;44(2):122-9. doi: 10.1159/000447019. Epub 2016 Aug 4. PMID 27487357